CLINICAL TRIAL: NCT00267696
Title: A Phase II Study of Gemcitabine/Carboplatin/Bevacizumab in Platinum Sensitive Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Patients.
Brief Title: Study of Gemcitabine/Carboplatin/Bevacizumab to Treat Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Larry Copeland, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-05070
Record Dates: First submitted 2005-12-19; First posted 2005-12-21 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: ovarian cancer; platinum sensitive cancer; fallopian tube cancer; peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine/carboplatin/bevacizumab (Experimental): A regimen consisting of gemcitabine(1000 mg/m2)/carboplatin(AUC 3) / bevacizumab(Avastin®)(10mg/kg) will be administered on day 1 and day 15 of a 28 day cycle.
  Interventions: Drug: Bevacizumab; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab(Avastin)=10mg/kg on day 1, day 15 of a 28 day cycle.
  Other Names: Avastin®
Drug: Gemcitabine — A regimen consisting of gemcitabine 1000 mg/m2 will be administered on day 1 and day 15 of a 28 day cycle
Drug: Carboplatin

SUMMARY:
The purpose of this study is to test the effectiveness, safety and tolerability of the drug combination: gemcitabine, carboplatin and bevacizumab in patients that have been diagnosed with platinum sensitive recurrent ovarian cancer, fallopian tube or primary peritoneal cancer.

DETAILED DESCRIPTION:
In this study participants will receive the drug combination gemcitabine/carboplatin and bevacizumab once every two weeks. As long as there is evidence that the tumor is not growing and the participant is not experiencing any unacceptable side effects, participation can continue up to 2 years. The study is being done to find the effectiveness, safety and tolerability of this combination of chemotherapy drugs. Bevacizumab affects the growth of new blood vessels in the body. It is part of this study to see if stopping the growth of new blood vessels in the body will help stop the growth and the spread of cancer. The other two chemotherapy drugs, gemcitabine and carboplatin, are currently being used together for the treatment of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the ovaries, fallopian tube or abdominal lining has come back after more than 6 months from the last platinum based chemotherapy treatment.
* Disease must be detected by CT or CA125 level must be elevated or cancerous ascites must be present.
* History of at least one therapy of platinum based chemotherapy.

Exclusion Criteria:

* Participation in another experimental drug study
* Heart disease or high blood pressure
* History of a stroke within the past 6 months
* Vascular disease, or bleeding problems
* Brain cancer
* Major Surgical Procedure within 28 days prior to start date
* Minor surgical procedures within 7 days prior to start date
* Pregnant or lactating
* Abdominal or bowel problems like bleeding
* History of abdominal fistula, GI perforation or Intra-abdominal abscess
* Serious, non-healing wound, ulcer or bone fracture
* Acute hepatitis
* Active infections requiring antibiotics
* Inability to comply with study or follow up procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-11; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry J. Copeland, MD, Principal Investigator — Professor & Chair Department of Obstetrics & Gynecology and Division of Gynecologic Oncology
Locations (1):
- The Ohio State University & James Cancer Hospital, Columbus, Ohio, United States

REFERENCES:
- [Result] Richardson DL, Backes FJ, Seamon LG, Zanagnolo V, O'Malley DM, Cohn DE, Fowler JM, Copeland LJ. Combination gemcitabine, platinum, and bevacizumab for the treatment of recurrent ovarian cancer. Gynecol Oncol. 2008 Dec;111(3):461-6. doi: 10.1016/j.ygyno.2008.08.011. Epub 2008 Sep 30. PMID 18829088
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2006 through August 2010
Groups:
- Gemcitabine/Carboplatin/Bevacizumab: A regimen consisting of gemcitabine(1000 mg/m2)/carboplatin(AUC 3) / bevacizumab(Avastin®)(10mg/kg) will be administered on day 1 and day 15 of a 28 day cycle.
  Bevacizumab: Bevacizumab(Avastin)=10mg/kg on day 1, day 15 of a 28 day cycle.
  Gemcitabine: A regimen consisting of gemcitabine 1000 mg/m2 will be administered on day 1 and day 15 of a 28 day cycle
  Carboplatin
Period: Overall Study
Arm/Group | Gemcitabine/Carboplatin/Bevacizumab
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine/Carboplatin/Bevacizumab: A regimen consisting of gemcitabine(1000 mg/m2)/carboplatin(AUC 3) / bevacizumab(Avastin®)(10mg/kg) will be administered on day 1 and day 15 of a 28 day cycle.
  Bevacizumab: Bevacizumab(Avastin)=10mg/kg on day 1, day 15 of a 28 day cycle.
  Gemcitabine: A regimen consisting of gemcitabine 1000 mg/m2 will be administred on day 1 and day 15 of a 28 day cycle
  Carboplatin
Arm/Group | Gemcitabine/Carboplatin/Bevacizumab
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 60.0 [42.0 to 77.0]
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 36
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: patients]
  United States | 45
ECOG (Eastern Cooperative Oncology Group) Performance Status [Number; unit: patients]
  0 (Fully active) | 34
  1 (Restricted in physical activity) | 11
Primary disease site [Number; unit: patients]
  Ovarian | 40
  Primary peritoneal | 4
  Tubal | 1
Primary disease stage [Number; unit: patients]
  Stage 1-2 (cancer located in ovaries or pelvis) | 7
  Stage 3 (cancer in ovaries spread to peritoneum) | 34
  Stage 4 (cancer has spread to distant organs) | 4
Primary disease grade [Number; unit: patients]
  G2(tissue moderately differentiated) | 3
  G3(tissue poorly differentiated/undifferentiated) | 42
Platinum-free interval [Median (Full Range); unit: months] | 15 [6 to 125]
Disease status at study enrollment [Number; unit: patients]
  Measurable disease | 33
  Non-measurable disease (CA125) | 12

OUTCOME MEASURES:

1. Primary Outcome: Determine the Antitumor Activity of Gemcitabine/Carboplatin/Bevacizumab Regimen as Measured by the Probability of Surviving Progression-free for at Least 6 Months or Responding.
Description: Progression-free survival (PFS) by RECIST, and safety. RECIST verison 1.0 was used for the assessment of progression and was based on radiologic evaluation.
Time Frame: up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine/Carboplatin/Bevacizumab
Number analyzed (Participants) | 45
months | 13.3 [11.3 to 15.3]

2. Secondary Outcome: Overall Survival for Patients Treated With the Regimen.
Description: The period of time from study entry until disease progression or date of last contact.
Time Frame: To progression of Disease
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine/Carboplatin/Bevacizumab
Number analyzed (Participants) | 45
months | 36.1 [26.7 to 45.5]

ADVERSE EVENTS:
Time Frame: Toxicity was graded according to the CTCAE-3. Patients were observed for adverse events fro 30 days after treatment discontinuation, and for survival every 3 months until death.
Arm/Group | Gemcitabine/Carboplatin/Bevacizumab
Serious Adverse Events (participants affected / at risk) | 4/45
Other Adverse Events (participants affected / at risk) | 39/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Carboplatin/Bevacizumab (N=45)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Cerebrovascular events (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Carboplatin/Bevacizumab (N=45)
Hematologic (Blood and lymphatic system disorders) | 39 (39) — Grade 3 and 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No